CLINICAL TRIAL: NCT05273593
Title: Confocal Laser Endomicroscopy During TransUrethral Resection for Improving Bladder Cancer Diagnosis and Treatment
Brief Title: Confocal Laser Endomicroscopy During TransUrethral Resection for Improving BC Diagnosis and Treatment
Acronym: CLETUR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Prof.dr. H.P. Beerlage, Head of Department of Urology, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL71360.018.19
Record Dates: First submitted 2020-03-19; First posted 2022-03-10 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Bladder Cancer; CLE
Keywords: Confocal Laser Endomicroscopy; CLE; Bladder cancer; Diagnosis; Imaging techniques
MeSH Terms: conditions — Urinary Bladder Neoplasms; Disease

STUDY DESIGN:
Intervention Model Description: Feasibility study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Confocal Laser Endomicroscopy (CLE) — Administration of fluorescein, intravesically and intravenously. CLE measurements with flexible and rigid probe of papillary bladder tumour and rigid probe-measurement of resection bed.

SUMMARY:
A prospective monocenter diagnostic accuracy study of Confocal Laser Endomicroscopy (CLE) for Bladder Cancer(BC) to assess two primary objectives:

1. The diagnostic accuracy of flexible probe-based confocal laser endomicroscopy (CLE) compared to histopathology of the resection specimen.
2. The diagnostic accuracy of CLE-based assessment of the surgical radicality of the resection bed (radical vs irradical) in comparison with histopathology of a biopsy of the resection bed.

All patients with a papillary bladder tumor on cystoscopy will be included in this trial.

DETAILED DESCRIPTION:
Rationale:

Initial evaluation of gross hematuria consists of White Light Cystoscopy (WLC). Urine cytology combined with contrast imaging of the upper urothelial tract is performed when a bladder tumor is seen. Follow up of non-muscle invasive bladder carcinoma (NMIBC) after initial treatment consists of similar steps. When a suspected lesion is visualized, a transurethral resection of the bladder tumor (TURBT) is performed for therapeutic and diagnostic purposes. TURBT is considered to be the gold standard for diagnosis of urothelial carcinoma of the bladder (UCB). High recurrence rates of UCB after TURBT are reported, leading to repetitive surgery and high costs. In certain cases of high grade UCB a second look TURBT has proven to be beneficial after primary resection to ensure radical resection. Furthermore, recent research suggests that active surveillance for low-grade bladder tumors is safe. Confocal laser endomicroscopy (CLE), a high resolution optical imaging technique that can be used in combination with endo-urological procedures, seems promising to improve diagnosis of urothelial cancer, possibly without the need for immediate transurethral resection to obtain histological confirmation. CLE characteristics of UCB have been determined and validated using rigid probes, which are incompatible with flexible cystoscopes used for outpatient cystoscopies. With the present study, we aim to assess the diagnostic value of flexible probe based CLE for diagnosis and grading of UCB. Furthermore to possibly prevent second look TURBT in the future,an assessment of CLE features of the resection bed using a rigid CLE-probe will be performed.

Objective:

Primary objectives:

This study is two-fold and, therefore, has two primary objectives:

1. Investigating the diagnostic accuracy of CLE (Cystoflex™F probe) during flexible cystoscopy for diagnosis and grading of urothelial carcinoma of the bladder.
2. To investigate the diagnostic potential of CLE (Cystoflex™ UHD-R probe) for the assessment of the surgical radicality after transurethral resection of a bladder tumor (after TURBT)

Secondary objective:

- To construct a convolutional neural network for computer aided assessment of CLE images for diagnosis and grading of UCB.

Study design:

This is a prospective monocenter, observational diagnostic accuracy study. Diagnostic accuracy study to compare the CLE-based diagnosis with the histopathologic findings.

Study population: All patients >18 years old with a papillary bladder tumor who are planned for TURBT are eligible for this study. We will include 60 patients in this pilot study.

Intervention: At the operation theatre, before performing a TURBT for the standard clinical care, we introduce a flexible cystoscope to map the bladder, then we record CLE images of the index lesion using the Cystoflex™F. Subsequently, we replace the flexible scope by the (rigid) resectoscope. We acquire additional images with the Cystoflex™ UHD-R rigid probe. We perform the TURBT. After completion of the TURBT, we introduce the Cystoflex™ UHD-R probe again for imaging of the resection bed. At a later stage correlation with a standard biopsy of the resection bed will be performed.

For CLE imaging, a fluorescent contrast agent (fluorescein) will be used intravesically and intravenously, respectively, to temporarily stain the extracellular matrix of the urothelium. We will introduce fluorescein for intravesical use through a bladder catheter and rinse the fluorescein out of the bladder after an indwelling time of 5-10 minutes. Before CLE measurement of the resection bed we will administer fluorescein intravenously.

Main study parameters/endpoints:

1. Overall accuracy, sensitivity and specificity of flexible probe CLE-based diagnosis (benign vs malignant) and grading (low-grade versus high-grade) in comparison with the histopathology of the resection specimen.
2. Overall accuracy, sensitivity and specificity of CLE-based assessment of the surgical radicality of the resection bed (radical versus irradical) in comparison with the histopathology of the biopsy of the resection bed.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Participants will not benefit directly from this study. We hypothesize, however, that the results of this study will contribute to improvements in the diagnostic and surgical procedure for UCB. Outpatient-based cystoscopy with the potential diagnostic certainty of CLE-based grade assessment may enable active surveillance in low-risk UCB, and thus may even lead to a reduction in surgical procedures. We will introduce a CLE probe before TURBT via the working channel of the flexible cystoscope and hold it in direct contact with the bladder tumor to obtain CLE images. Before image acquisition of the bladder tumor we administer fluorescein intravesical, which is a fluorescent dye, used regularly intravenously in ophthalmatology. Before image acquisition of the resection bed we administer fluorescein intravenously. In patients not known with an allergy to this dye, this is a safe procedure. Patients with a known allergic reaction to fluorescein cannot participate in this study. Patients will be exposed to approximately 20 minutes of extra surgery time and the introduction of a flexible cystoscope compared to regular TURBT. As a result there is little burden to study participation for the patients. Adverse events are not expected based on previous experiences. The hospital's internal protocol for standard clinical care and histopathologic evaluation are not going to be affected by the study protocol.

ELIGIBILITY:
Inclusion Criteria:

* Display a papillary bladder tumor on cystoscopy.
* >18 years of age.
* Has given written informed consent.

Exclusion Criteria:

* Patients with a known allergy to fluorescein.
* Pregnancy or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2021-11-12 (Actual); Study Completion 2021-11-12 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of flexible-probe based CLE(pCLE) for the diagnosis of urothelial carcinoma of the bladder (UCB) | Consensus panel within 12 months of start of study.
  Diagnostic accuracy (sensitivity, specificity, negative predictive value and positive predictive value) of flexible probe based CLE for the diagnosis (low-grade malignant, high-grade malignant) of urothelial carcinoma of the bladder.
Diagnostic potential of probe based CLE for assessment of surgical radicality after transurethral resection of a bladder tumour (TURBT). | Consensus panel within 12 months of start of study.
  To investigate the diagnostic potential of CLE for the assessment of the surgical radicality (residual tumor/no residual tumor) after TURBT.
Diagnostic potential of probe based CLE for assessment of depth of resection after transurethral resection of a bladder tumour (TURBT). | Consensus panel within 12 months of start of study.
  To investigate the diagnostic potential of CLE for depth of resection (according to the tissue in the resection margin: urothelium, submucosa, m. detrusor or perivesical fatty tissue) after TURBT.

SECONDARY OUTCOMES:
Computer aided assessment of pCLE images for diagnosis and grading of UCB | Within 24 months after starting study
  To construct a convolutional neural network for computer aided assessment of pCLE images for diagnosis and grading of UCB.

CONTACTS AND LOCATIONS:
Overall Officials: J. R. Oddens, MD, PhD, Principal Investigator — Staff member of Urology Department
Locations (1):
- Academic Medical Center, Amsterdam, North Holland, Netherlands